CLINICAL TRIAL: NCT04249570
Title: Efficacy of Gastrostomy Tube Coated With Povidone-iodine for Reducing Peristomal Infection Rate After PEG Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V103A-012
Record Dates: First submitted 2014-11-25; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Infection
Keywords: percutaneous endoscopic gastrostomy; Povidone-iodine; peristomal infection
MeSH Terms: conditions — Infections | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodine (Experimental): gastrostomy feeding tube is coated with a layer of Betadine by aseptic gauze before PEG technique
  Interventions: Other: Povidone iodine
- No iodine (No Intervention): gastrostomy feeding tube is not coated with a layer of Betadine by aseptic gauze before PEG technique

INTERVENTIONS:
Other: Povidone iodine
  Other Names: Betadine
  Arms: Iodine

SUMMARY:
Percutaneous endoscopic gastrostomy (PEG) was created to replace surgical gastrostomy in patients who are needed long-term tube feeding. PEG has less severe complication rate or mortality rate compared with traditional surgical gastrostomy. However, there are still some mild complications which cannot be completely prevented and peristomal infection is the most common one. Povidone-iodine (PVP-I) exhibits broad range of microbicidal activity via increasing the solubility of iodine. In our study, the gastrostomy feeding tube will be coated with a layer of Betadine before PEG technique.

Investigators expect gastrostomy feeding tube coated with Betadine will reduce the oropharyngeal, esophageal and gastric bacteria colonization rate, followed by reducing peristomal infection rate.

DETAILED DESCRIPTION:
Percutaneous endoscopic gastrostomy (PEG), or placement of a gastrostomy tube with the aid of an endoscope, was first reported by a pediatrist in 1980. It was created to replace surgical gastrostomy and used widely in patients who are needed long-term tube feeding. There are three kinds of PEG techniques, including pull method, push method and introducer method. Among them, pull method is the most widely accepted technique due to its simplicity of insertion.

PEG has less severe complication rate or mortality rate compared with traditional surgical gastrostomy. However, there are still some mild complications which cannot be completely prevented and peristomal infection is the most common one. The major cause of peristomal infection is that oropharyngeal bacteria colonized gastrostomy feeding tube while undergoing PEG placement with pull method or push method, then bacteria was brought to the stoma via gastrostomy feeding tube and induced peristomal infection.

Povidone-iodine (PVP-I) is a stable chemical complex of polyvinylpyrrolidone (povidone, PVP) and iodine. It exhibits broad range of microbicidal activity via increasing the solubility of iodine. A retrospective study in Japan demonstrated that using Povidone-iodine gargling solution before PEG technique reduced peristomal infection rate. Besides, many studies demonstrated that gingival degerming by Povidone-iodine irrigation prior to extraction or gingivectomy reduced the oral bacterial colonies and postoperative infection rate.

The investigators will use Betadine (10% Povidone iodine) as experimental drug. The gastrostomy feeding tube will be coated with a layer of Betadine by aseptic gauze before PEG technique. Investigators expect that gastrostomy feeding tube coated with Betadine will reduce the oropharyngeal, esophageal and gastric bacteria colonization rate, followed by reducing peristomal infection rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with central nervous system disorder, head and neck cancer, esophageal motility disorder or swallowing dysfunction related to face trauma, who are the candidates for percutaneous endoscopic gastrostomy under doctors' suggestion
* Patients between 20 and 100 years old

Exclusion Criteria:

* History of upper abdominal surgery
* Intra-abdominal hemorrhage
* Massive ascites
* Severe coagulopathy
* Malignancy infiltration to the stomach
* Severe left lobe hypertrophy of liver
* High position of transverse colon
* Esophageal stricture
* Thyroid disease
* Allergy to Cephalosporin or Povidine iodine
* Current antibiotics use or use antibiotics in recent 2 days

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Peristomal infection rate | two weeks
  For each patient, the peristomal area was evaluated daily for 2 weeks after PEG placement. The presence of erythema and of exudate were scored on a scale of 0 to 4; induration was scored on a scale of 0 to 3. Criteria for infection were a maximum combined score of 8 or higher, or the presence of microscopic and microbiologic evidence of suppurating exudate.

SECONDARY OUTCOMES:
Pneumonia | two weeks
  Diagnosis of aspiration pneumonia after PEG with clinical, biological and radiological :criteria including fever, leucocytes, broncho alveolar secretion, chest radiography and bacteriological identification.
Serum CRP level changes before and after PEG placement | 3 days
  Serum CRP level was check before and after PEG placement. The timing was early morning at procedure day and early morning on the next day.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Hou, MD, Principal Investigator — Department of Gastroenterology, Taipei Veterans General Hospital, Taipei, Taiwan; Yen-Po Wang, Study Director — Endoscopy Center for Diagnosis and Treatment, Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taiwan, Taipei, Taiwan

REFERENCES:
- [Derived] Chen YJ, Hou MC, Yang TC, Lee PC, Wang YP, Huang YH, Lee FY. Effectiveness of betadine-coating gastrostomy tube to reduce peristomal infection after percutaneous endoscopic gastrostomy: a randomized controlled trial. BMC Gastroenterol. 2023 May 15;23(1):155. doi: 10.1186/s12876-023-02702-w. PMID 37189057